CLINICAL TRIAL: NCT05720780
Title: Can Rehabilitation Training With Music-support Increase Exercise Tolerance in Individuals With COPD and CRF Compared to Rehabilitation Training Alone? A Randomized Control Trial.
Brief Title: Rehabilitation Training With Music-support & Exercise Tolerance in COPD and CRF Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICS Maugeri 2712 CE
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: COPD
Keywords: distracting auditory stimulus (DAS); COPD; CRF; music therapy; rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual training with the support of music (MS) (Experimental): This is the group performing training with the support of the music; it will be the intervention study group (MS)
  Interventions: Other: MS group
- Usual training without music (C) (Active Comparator): This is the usual training group without the support of the music, it will be the control group (C)
  Interventions: Other: C group

INTERVENTIONS:
Other: MS group — All patients will perform the usual training by listening a piece of music of the same duration as the training. The patient will be able to choose among 4 different musical proposals corresponding to 4 different styles: rock, modern, jazz and classical. The song chosen by the patient will be the musical support for all the sessions of training on the cycle ergometer. The musical pieces will be composed with a constant rhythm (bpm=60) which, from a tonal point of view, will echo the pedaling movement. The constant rhythm will be superimposed on musical patterns in the form of loops in the styles mentioned. The musical support will assume a "priming" (activation) and "dragging" (synchronization) function, facilitating movement planning/synchronization and creating a pleasant context in which to carry out training
  Other Names: Experimental
  Arms: Usual training with the support of music (MS)
Other: C group — All patients will perform 12 to 14 supervised sessions depending on the center they belong to (5-6 sessions/week) each consisting of 30 minutes of exercise at the cycle ergometer plus 3 minutes of warm-up and 3 minutes of recovery. After a warm-up phase at 0 W, the initial workload will be set to 60% of the theoretical maximum. Intensity increases or decreases of 10 W will be made according to the criteria of Maltais et al (workload will be increased when patients will report dyspnea and/or leg fatigue as ≤3 on a Borg scale modified to 10 points of perceived effort. The training load will remain unchanged if the Borg score is 4 or 5 and will be reduced for scores ≥6). Patients will have to maintain a pedaling frequency between 55 and 60 rpm.
  Other Names: Active Comparatore
  Arms: Usual training without music (C)

SUMMARY:
Therapeutic-rehabilitative interventions supported by music can be considered important resources in many clinical contexts. Some studies report the improvement of psychological (i.e. anxiety) and physiological parameters such for example, dyspnea, blood pressure, quality of life, sleep disturbances, etc. through voice, singing, exercise with wind instruments, and sometimes listening to music. Among the various instruments proposed to support the physical training of COPD patients, music was also tested and, in particular, music as a distracting auditory stimulus (DAS) has been used to increase exercise and physical activity adherence and to reduce the perception of dyspnea in COPD subjects.

This randomized controlled trial will compare -in patients with COPD and CRF- the effects of the addiction of music to the training on exercise capacity (possible improvement of endurance and reduction of fatigue and dyspnea) with respect to the usual rehabilitation modality (no music).

DETAILED DESCRIPTION:
Background:

Several studies had proposed to support the physical training of COPD patients with and without chronic respiratory failure (CRF), with external systems such as oxygen therapy, high-flow oxygen therapy, and noninvasive ventilation, to improve performance during exercise training.

More recently, the role of music therapy has been also tested. Therapeutic-rehabilitative interventions supported by music can be considered important resources in many clinical contexts. The active and receptive approaches of music therapy (based respectively on sound-music interaction with the patient and introspection through musical listening techniques) are intended to improve relationships in terms of communication, expression, and regulation of emotions. Anyway, the use of sound and music is widely used in the rehabilitation context: music therapy in the neurological field, for example, consists of about 20 techniques that aim to improve neuromotor, and cognitive and sensory rehabilitation, as well. Some studies report the improvement of psychological (anxiety) and physiological parameters such as, for example, dyspnea, blood pressure, quality of life, sleep disturbances, etc. through voice, singing, exercise with wind instruments, and sometimes listening to music. OIn the studies conducted on patients with COPD, listening to music-staff during an exercise training session, have shown greater tolerance to high-intensity exercise demonstrated by a greater endurance time as well as listening to rhythmic music has allowed for greater exercise intensity. Furthermore, music as a distracting auditory stimulus (DAS) has been used to increase exercise and physical activity adherence and to reduce the perception of dyspnea in COPD subjects. A review of thirteen studies using DAS in 415 participants demonstrated that DAS increased exercise capacity when applied for at least 2 months of training (in most cases during walking), while the quality of life improved only after training of at least 3 months; the patient had less dyspnea using DAS during exercise, but this was not consistently observed in short-term exercise tests or the symptom management strategy at rest.

To date, there are no studies that evaluate whether a medium-term training cycle supported by music can further improve exercise tolerance in deconditioned subjects, such as patients with COPD and chronic respiratory failure (CRI), in comparison to subjects performing training without music.

In the present study, music will therefore be used to support training in a group of randomized patients with COPD and CRF to improve their endurance and reduce the perception of fatigue and dyspnea with respect to patients performing the usual rehabilitation training (without music). Possible improvements in performance and related physiological parameters are expected.

Methods:

This is a multicenter RCT study with a low-risk intervention. Patients with a diagnosis of COPD, according to the Global Initiative for Lung Disease (GOLD) criteria, will be recruited for this purpose and randomly assigned to two groups: training without music (C) and training with the addition of music (MS). A single list of randomization (1:1 randomization ratio in fixed blocks of 4 (https://www.randomizer.org/) will be created by a person external to the healthcare staff.

The treatment in the two groups is reported in the intervention section. All training sessions will be supervised by a physiotherapist and the only difference between the two groups will be the music listening in the MS group other than training.

At baseline (the date of randomization), the investigators will collect clinical evaluations as follows:

* Demographic and anthropometric data
* Post-bronchodilator spirometry and plethysmography (Forced Expiratory Volume at 1 second, Forced Vital Capacity, Residual Volume, Inspiratory Capacity). The results will be expressed as absolute values and percentages of the predicted values according to Quanjer.
* Cumulative Illness Rating Score (CIRS)

At baseline and the end of the rehabilitation program, the investigators will collect:

* 6-minute walk test (6MWT): Borg fatigue and dyspnea scores and pulse oximetry (SpO2) will be recorded at the beginning and end of the test. The distance walked in meters, as well as the SpO2 nadir and the SpO2/heart rate (HR) ratio will be recorded at the end of the test;
* Respiratory muscle strength will be evaluated through the maximum inspiratory pressures (MIP) and expiratory pressures (MEP) using an electronic pressure gauge (Precision Medical, Northampton, PA, USA);
* Strength of quadriceps muscles will be evaluated with a handheld dynamometer (Chatillon X-3328 Series; AMETEK, Inc, Berwyn, PA, USA). The maximum voluntary contraction will be expressed in kilograms;
* Arterial blood gases will be evaluated on blood samples taken from the radial artery while patients, seated, breathe room air (PaO2, PaCO2, pH).
* Exercise capacity will be assessed with a Constant Load Exercise Test (CLET) on a cycle ergometer. The workload will be set at 80% of the maximum workload expected by the 6MWT performed at baseline. Heart rate, saturation, blood pressure, Borg dyspnea and Borg fatigue evaluations will be recorded and tabulated at the end of each minute of the test.

At the beginning of each training session (T start) and at the end of each training session (T end) the following information will be collected:

* Heart rate,
* oxygen saturation (satO2),
* dyspnea and muscle fatigue measured with a BORG scale (0-10).

The reasons for drop-out will be defined as follows:

1. Unable to sustain at least 12 sessions of training;
2. Poor adherence due to psychological and personal problems during training (self-discharge, personal commitment);
3. Exacerbation of COPD/pneumonia;
4. Acute events with or without premature hospital discharge;
5. Protocol or device rejection The Outcome measures are reported in the dedicated section. The statistical evaluation will be conducted with the STATA 11 program (StataCorp LLC). Continuous variables will be expressed as mean and standard deviation (or median and quartiles) while categorical or binary variables as a percentage.

The sample size will be calculated on the percentage of patients who will be able to achieve the MCID (Minimal Clinical Important Difference) of 30 meters at 6MWT in COPD (responders), using a frequency comparison test for independent samples (chi-square) with a = 0.05, b= 0.80. Estimating that the number of improving patients (responders) in the control group is equal to 63% while in the study group 83%, the estimated sample is 156 patients (78 per group). Therefore, 26 patients per center are assumed.

The estimation of 63% in the control group derives from a previous work on the effect of addiction of high oxygen flows during training in a similar population; while the estimation of the proportion of improvers in the study group is based on data on the time of performance with the use of music (+19%) in patients in "an acute phase of disease".

Secondary analyses will be performed using appropriate parametric and non-parametric tests to verify differences between groups in response to treatment (T-test or Wilcoxon to evaluate the difference between means or medians and chi-square test to evaluate the difference between frequencies). A secondary evaluation by logistic regression will also be performed to verify the baseline characteristics predictive of improvement in responders. A p-value <.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (Forced expiratory volume in 1 second / post-bronchodilator forced vital capacity < 0.7) without functional reversibility
* Chronic respiratory failure with stable hypoxia (PaO2 < 60 mmHg in room air)
* Long Term Oxygen Therapy (LTOT) for at least 3 months
* Clinical stability: pH range 7.38-7.42, with no recent exacerbations in the last 7 days and no changes in drug therapy in the previous 7 days

Exclusion Criteria:

* Non-invasive ventilation at home
* Cognitive impairment (Mini-Mental State Examination Score < 22)
* Asthma or evidence of bronchodilator response
* Pulmonary fibrosis
* Obstructive sleep apnea syndrome
* Lung cancer
* Active microbial infections
* Neuromuscular, orthopedic, and/or medical conditions that preclude testing
* Pulmonary rehabilitation program in the previous 6 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in effort tolerance at 6 minutes walking test: Minimal Clinical Important Difference (MCID) at 6MWT | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to usual training (without music), is more effective in improving the exercise capacity measured in terms of the number of patients able to achieve the MCID (Minimal Clinical Important Difference) of 30 meters at the six-minute walking test (6MWT).

SECONDARY OUTCOMES:
Change in effort tolerance at 6 minutes walking test: distance at 6MWT | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to a usual training (without music), is more effective in improving the exercise capacity measured in terms of meters covered in six minutes
Change in effort tolerance at the constant load exercise test (CLET) | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to a usual training (without music), is more effective in improving the exercise capacity measured in terms of time measured in seconds at the CLET
Change in dyspnea: total sessions | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to a usual training (without music), is more effective in reducing dyspnoea (measured with the Borg scale) during training (total sessions)
Change in dyspnea:iso-times at CLET | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to a usual training (without music), is more effective in reducing dyspnea at the CLET by evaluating dyspnea at the same minutes observed in the initial test (iso-times)
Change in dyspnea during daily life activities (ADL) by Medical Research Council (MRC) | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to usual training (without music), is more effective in reducing dyspnea during ADL measured with MRC. We will evaluate Dyspnoea in activities of daily life through the modified Medical Research Council (mMRC) scale. The 1-5 stage scale is used alongside the questionnaire to establish clinical grades of breathlessness, where 0 is the best value and 4 is the worst value.
Change in dyspnea during daily life activities (ADL) by Barthel Dyspnea Index | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to a usual training (without music), is more effective in reducing dyspnea during ADL measured with Barthel Dyspnea Index.
  Dyspnoea assessment during ADLs based on BI items is described by the Italian version of Barthel index Dyspnea (BiD). BiD is a unique instrument able to measure both motor and respiratory disabilities. Scores range from 0 to 100, being 100 the worst value.
Change in the disease impact status by COPD Assessment Test (CAT) | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether the training exercise with music, compared to usual training (without music), is more effective in improving the disease impact status measured with CAT.
  Disease impact by the COPD assessment test (CAT). Range of CAT scores from 0 to 40. Higher scores denote a more severe impact of COPD on a patient's life. CAT scores from 21 to 30 indicate a high impact of COPD on the patient's life, as shown at admission. At discharge, the average CAT score turned out a medium impact, as a defined range from 10 to 20 points. The minimal clinically important difference (MCID) for CAT is supposed to be a change of 2 points.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Study Director — ICS Maugeri IRCCS, respiratory rehabilitation of the Institute of Lumezzane
Locations (6):
- Italy (6):
  - ICS Maugeri IRCCS, respiratory rehabilitation of the Institute of Telese, Telese Terme, Benevento
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Lumezzane, Lumezzane, Brescia
  - ICS Maugeri IRCCS, respiratory rehabilitation of the Institute of Montescano, Montescano, Pavia
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Tradate, Tradate, Varese
  - ICS Maugeri IRCCS, respiratory rehabilitation of the Institute of Bari, Bari
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Pavia, Pavia

REFERENCES:
- [Background] Lee AL, Desveaux L, Goldstein RS, Brooks D. Distractive Auditory Stimuli in the Form of Music in Individuals With COPD: A Systematic Review. Chest. 2015 Aug;148(2):417-429. doi: 10.1378/chest.14-2168. PMID 25741661
- [Background] Braun Janzen T, Koshimori Y, Richard NM, Thaut MH. Rhythm and Music-Based Interventions in Motor Rehabilitation: Current Evidence and Future Perspectives. Front Hum Neurosci. 2022 Jan 17;15:789467. doi: 10.3389/fnhum.2021.789467. eCollection 2021. PMID 35111007
- [Background] Canga B, Azoulay R, Raskin J, Loewy J. AIR: Advances in Respiration - Music therapy in the treatment of chronic pulmonary disease. Respir Med. 2015 Dec;109(12):1532-9. doi: 10.1016/j.rmed.2015.10.001. Epub 2015 Oct 19. PMID 26522499
- [Background] Ho CF, Maa SH, Shyu YI, Lai YT, Hung TC, Chen HC. Effectiveness of paced walking to music at home for patients with COPD. COPD. 2012 Aug;9(5):447-57. doi: 10.3109/15412555.2012.685664. Epub 2012 May 29. PMID 22643033
- [Background] Huang J, Yuan X, Zhang N, Qiu H, Chen X. Music Therapy in Adults With COPD. Respir Care. 2021 Mar;66(3):501-509. doi: 10.4187/respcare.07489. Epub 2020 Nov 3. PMID 33144384
- [Background] Kaasgaard M, Rasmussen DB, Andreasson KH, Hilberg O, Lokke A, Vuust P, Bodtger U. Use of Singing for Lung Health as an alternative training modality within pulmonary rehabilitation for COPD: a randomised controlled trial. Eur Respir J. 2022 May 19;59(5):2101142. doi: 10.1183/13993003.01142-2021. Print 2022 May. PMID 34625480
- [Background] Shingai K, Kanezaki M, Senjyu H. Distractive Auditory Stimuli Alleviate the Perception of Dyspnea Induced by Low-Intensity Exercise in Elderly Subjects With COPD. Respir Care. 2015 May;60(5):689-94. doi: 10.4187/respcare.03533. Epub 2015 Jan 13. PMID 25587171
- [Background] Lee AL, Dolmage TE, Rhim M, Goldstein RS, Brooks D. The Impact of Listening to Music During a High-Intensity Exercise Endurance Test in People With COPD. Chest. 2018 May;153(5):1134-1141. doi: 10.1016/j.chest.2017.12.001. Epub 2017 Dec 16. PMID 29253555
- [Background] Okamoto J, Furukawa Y, Kobinata N, Yoshikawa H, Araki F, Yagyu A, Iwasaka Y. Combined effect of pulmonary rehabilitation and music therapy in patients with chronic obstructive pulmonary disease. J Phys Ther Sci. 2021 Oct;33(10):779-783. doi: 10.1589/jpts.33.779. Epub 2021 Oct 13. PMID 34658524
- [Background] Panigrahi A, Sohani S, Amadi C, Joshi A. Role of music in the management of chronic obstructive pulmonary disease (COPD): a literature review. Technol Health Care. 2014;22(1):53-61. doi: 10.3233/THC-130773. PMID 24398814
- [Background] Raglio A, Oasi O. Music and health: what interventions for what results? Front Psychol. 2015 Mar 2;6:230. doi: 10.3389/fpsyg.2015.00230. eCollection 2015. No abstract available. PMID 25784891
- [Background] Raglio A. Music and neurorehabilitation: Yes, we can! Funct Neurol. 2018 Oct/Dec;33(4):173-174. No abstract available. PMID 30663962
- [Background] Vitacca M, Paneroni M, Zampogna E, Visca D, Carlucci A, Cirio S, Banfi P, Pappacoda G, Trianni L, Brogneri A, Belli S, Paracchini E, Aliani M, Spinelli V, Gigliotti F, Lanini B, Lazzeri M, Clini EM, Malovini A, Ambrosino N; Associazione Italiana Riabilitatori Insufficienza Respiratoria and Associazione Italiana Pneumologi Ospedalieri rehabilitation group. High-Flow Oxygen Therapy During Exercise Training in Patients With Chronic Obstructive Pulmonary Disease and Chronic Hypoxemia: A Multicenter Randomized Controlled Trial. Phys Ther. 2020 Aug 12;100(8):1249-1259. doi: 10.1093/ptj/pzaa076. PMID 32329780
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809